CLINICAL TRIAL: NCT03791970
Title: A Prospective, Single Center, Case-cohort Study Using the Orchid Drug Coated Balloon for Post-Dilatation of the Stent for Treatment of Long Lesions in Femoropopliteal Arteries
Brief Title: Stents Post-dilation With DCB or POBA in Femoropopliteal Arteries
Acronym: SFPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Kaichuang Ye, MD, PhD, Clinical Professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAL02
Record Dates: First submitted 2019-01-01; First posted 2019-01-03 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB for post-dilation (Experimental): DCB was used for post-dilation after stent placement. The DCB for post-dilation in this study is Orchid 035 DCB Catheter.
  Interventions: Device: Orchid 035 DCB Catheter
- POBA for post-dilation (Active Comparator): POBA was used for post-dilation after stent placement. POBA Catheter for post-dilation in this study can be Mustang, Dorado or others balloon catheters.
  Interventions: Device: POBA Catheter

INTERVENTIONS:
Device: Orchid 035 DCB Catheter — Stents placement for femoropopliteal arterial occlusions following with Orchid 035 DCB Catheter for post-dilation
  Arms: DCB for post-dilation
Device: POBA Catheter — Stents placement for femoropopliteal arterial occlusions following with POBA for post-dilation
  Arms: POBA for post-dilation

SUMMARY:
To compare the efficacy and safety of stent angioplasty with Orchid 035 Drug Coated Dilatation (DCB) and Plain Old Balloon Angioplasty (POBA) for post-dilatation for long (>10cm) femoropopliteal chronic total occlusion.

DETAILED DESCRIPTION:
A Prospective, Single Center, Case-cohort Study Using the Orchid Drug Coated Balloon for Post-Dilatation of the Stent for Treatment of Long Lesions in Femoropopliteal Arteries.

Patients will be selected based on the investigator's assessment, evaluation of the underlying disease and the eligibility criteria. The patient's medical condition should be stable, with no underlying medical condition which would prevent them from performing the required testing or from completing the study. Patients should also be geographically stable, willing and able to cooperate in this clinical study and remain available for long-term follow-up. A patient is considered enrolled in the study after obtaining the patients informed consent, if there is full compliance with the study eligibility criteria and after successful stent angioplasty for the occluded femoropopliteal arteries.

Prior to the index procedure the following tests and clinical data will be collected: informed consent for data collection, demographics, medical history, medication record, physical examination, clinical category of chronic limb ischemia (Rutherford category) and resting ankle-brachial index (ABI).

During the procedure, the vascular access can be achieved to the investigator's standard clinical practice. After successful lesion passage, diagnostic angiography of the lesion area and distal run-off is performed and angiographic measurements (vessel diameter, percentage stenosis and lesion length) are collected. All inflow-limiting lesion will be treated according to the investigators standard clinical practice before treatment of the target lesion. The study compares the efficacy and safety of stent angioplasty with Orchid 035 Drug Coated Dilatation (DCB) and Plain Old Balloon Angioplasty (POBA) for post-dilatation for long (>10cm) femoropopliteal chronic total occlusion. The indication for stent placement is based on the investigator's assessment. An expected total of 180 patients will be treated in the scope of this study. The lesion is located within the native superficial femoral artery and/or the popliteal artery. Prior to stents placement, pre-dilatation with the POBA balloon is mandatory. After stents placement, post-dilatation with the Orchid 035 DCB or POBA need to be performed. Patients will be invited for a follow-up visit at 1, 6 and 12 month post-procedure. The primary efficacy endpoint of the study is defined as the freedom from clinically-driven target lesion revascularization (TLR) at 12 months. Secondary endpoints include primary patency rate at 6 and 12 months, freedom from clinically-driven TLR at 6 months, clinical success at 1, 6 and 12 months and freedom from serious adverse events at pre-discharge, 1, 6 and 12 months follow-up.No other adjunctive therapies (atherectomy, laser) are allowed. The complete femoropopliteal vasculature should be treated in one single session, staged interventions are not allowed. All outflow-limiting lesions must be treated according to the hospital treatment standard.

The regular follow-ups are necessary to monitor the condition of the patient and the procedure. Patients will be invited for a follow-up visit at 1, 6 and 12 months after the index procedure. The following data will be collected during these follow-up visit: medication record, physical examination, rutherford categorization, ABI and color flow doppler ultrasound.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. The subject is legally competent and able to understand the information on the study, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions, and has duly signed the Informed Consent Form (ICF);
3. Rutherford Category 2-4;
4. Target de novo lesion(s) or non-stented restenotic lesion(s) has angiographic evidence of long-term occlusion (by visual estimate ≥10cm) and is amenable to treatment with stents placement;
5. Patients must be able to be treated with DCB or POBA for post-dilation;
6. Target vessel reference diameter is 4.0-7.0 mm (by visual estimate) and able to be treated with available device size matrix;
7. At least one patent native outflow artery to the ankle free from significant lesion (≥50% stenosis) as confirmed by angiography (treatment of outflow disease is NOT permitted; treatment of in-flow disease is permitted prior to treatment with stents placement).
8. No other prior vascular interventions (including contralateral limb) within 2 weeks before and/or planned 30 days after the protocol treatment, with the exception of remote common femoral patch angioplasty separated by at least 2 cm from the target lesion;
9. Female subjects of childbearing potential have a negative urine or serum pregnancy test within 7 days prior to index procedure;
10. Lesion location starts ≥1 cm below the common femoral bifurcation and P1 popliteal artery.

Exclusion Criteria:

1. Pregnant, lactating, or planning on becoming pregnant or men intending to father children;
2. Contraindication to stent or DCB or POBA per current information for use (IFU);
3. Life expectancy of <1 year;
4. Inability to take required antiplatelet/anticoagulant medications, or known contraindication (including allergic reaction) or sensitivity to contrast media, nickel, titanium or tantalum that cannot be adequately managed with pre- and post-procedure medication;
5. Intended treatment of outflow disease during the index procedure;
6. Intended use of laser, atherectomy or cryoplasty during index procedure;
7. Sudden symptom onset, acute vessel occlusion, or acute or subacute thrombus in target vessel;
8. History of stroke within 3 months;
9. History of myocardial infarction, thrombolysis or angina within 2 weeks of enrollment;
10. Participation in an investigational drug or another investigational device study until this study's primary endpoint is reached or previous enrollment in this study;
11. Another medical condition, which, in the opinion of the Investigator, may cause the patient to be noncompliant with the Concern/Information Need/Participation Willingness (CIP) or confound data interpretation;
12. Target vessel and/or lesion involves a previously placed stent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate | 12 months post-procedure
  Absence of a hemodynamically significant stenosis on duplex ultrasound (systolic velocity ratio no greater than 2.5) at the target lesion and without TLR

SECONDARY OUTCOMES:
Freedom from clinically-driven TLR | 6 and 12 months post-procedure
  TLR defined as a repeated intervention to maintain or re-establish patency within the region of the treated arteries

CONTACTS AND LOCATIONS:
Overall Officials: Xinwu Lu, MD, PhD, Study Chair — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (3):
- China (3):
  - Kaichuang Ye, Shanghai, Shanghai Municipality
  - Minyi Yin, Shanghai, Shanghai Municipality
  - Xiaobing Liu, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No